CLINICAL TRIAL: NCT06951126
Title: CT Prediction for Transcatheter Tricuspid Interventions
Acronym: CESAR-TR
Status: Recruiting | Type: Observational
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other); University Hospital Schleswig-Holstein (Other); University of Cologne (Other); Heart Center Leipzig - University Hospital (Other); Charite University, Berlin, Germany (Other); University of Bern (Other); University Medical Center Mainz (Other)
Responsible Party: Principal Investigator, Johannes Kirchner, Dr. med., Heart and Diabetes Center North-Rhine Westfalia
Other Study IDs: HDZ-KA CESAR-TR
Record Dates: First submitted 2025-04-16; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Tricuspid Regurgitation; Computed Tomography
Keywords: transcatheter tricuspid valve intervention; TTVI; TR; MSCT; Tricuspid regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study is to enhance the predictability of therapeutic success in transcatheter tricuspid valve intervention (TTVI) for patients with severe tricuspid regurgitation (TR). This will be achieved through automated analyses of pre-interventional computed tomography (CT) scans.

Severe tricuspid regurgitation is associated with poor patient outcomes. In advanced stages, pharmacological therapy becomes ineffective, and surgical intervention carries a high mortality risk. Given this clinical challenge, catheter-based treatment of the tricuspid valve has become a focal point of research.

One well-established treatment strategy is percutaneous tricuspid valve intervention, which aims to reduce regurgitation either through annuloplasty, leaflet-based edge-to-edge repair or valve replacement. This approach has been shown to significantly decrease the severity of regurgitation, leading to a dramatic reduction in symptom burden and a marked improvement in quality of life.

However, predicting which patients will benefit most from TTVI and determining the optimal technique for each individual remain largely unresolved challenges.

Artificial intelligence (AI)-powered software, such as heart.ai by LARALAB (Munich), enables automated measurement of anatomical structures captured via CT imaging. This technology already allows for rapid and precise assessment of cardiac chambers and the tricuspid annulus throughout the entire cardiac cycle, facilitating a comprehensive three-dimensional evaluation of right heart anatomy.

To refine patient selection and optimize procedural strategies for TR treatment, the researcher work a multi-center collaboration to analyze treatment outcomes and patient response to specific therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria:

* the patient underwent full cycle cardiac computed tomography for analysis of valvular heart disease
* a transcatheter tricuspid valve intervention is performed
* the patient is 18 years or older

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study includes patients with >moderate tricuspid regurgitation who underwent cardiac computed tomography and transcatheter tricupid valve intervention.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | 1 year
  Detection of mortality after transcatheter tricuspid intervention

SECONDARY OUTCOMES:
Residual Tricuspid Regurgitation | At discharge, 30 days and 1 year
  Grade of residual tricuspid regurgitation after transcatheter tricuspid valve intervention
rehospitalization rate | 1 year
  Detection of rehospitalization rate after transcatheter tricuspid intervention
reintervention rate | 1 year
  Detection of reintervention rate on the tricuspid valve after transcatheter tricuspid intervention
NYHA Class | 30 days and 1 year
  Changes on New York Heart Association functional class after transceather tricuspid valve intervention
Intraprocedural success | 30 days
  All of the following must be present:
  1. Absence of intraprocedural mortality or stroke; and
  2. Successful access, delivery, and retrieval of the device delivery system; and
  3. Successful deployment and correct positioning of the intended device(s) without requiring implantation of unplanned additional devices; and
  4. Adequate performance of the transcatheter device. Performance of devices whose purpose is a reduction in TR, should include the absence of tricuspid stenosis, reduction of total tricuspid regurgitation to optimal
  5. Absence of device-related obstruction of forward flow
  6. Absence of device-related pulmonary embolism
  7. Freedom from emergency surgery or reintervention during the first 24 h related to the device or access procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Herz- und Diabeteszentrum, Bad Oeynhausen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No